CLINICAL TRIAL: NCT02476747
Title: Comparison of Efficacy Between Cold Snare Polypectomy and Endoscopic Mucosal Resection in Treatment of Small Polyp
Brief Title: Cold Snare Polypectomy Versus. Endoscopic Mucosal Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Sik Byeon, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-0565
Record Dates: First submitted 2015-06-17; First posted 2015-06-19 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Colonic Polyp
Keywords: Colonic polyp
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cold snare polypectomy (Experimental): CSP will be performed by closing the snare loop after positioning the open snare at the point of lesion.
  Interventions: Other: CSP
- Endoscopic mucosal resection (Active Comparator): EMR will be performed in the way of drawing the lesion into the loop of the snare and resecting followed by saline injection to the its margin.
  Interventions: Other: EMR

INTERVENTIONS:
Other: EMR — performing EMR for patients with small polyp
  Arms: Endoscopic mucosal resection
Other: CSP — performing CSP for patients with small polyp
  Arms: Cold snare polypectomy

SUMMARY:
The investigators will investigate the efficacy of EMR compared to CSP in treatment of small colon polp (6~10mm).

One aim of this study was to investigate the necessity of EMR on resection of small colon polyp.

DETAILED DESCRIPTION:
With sized polyp from 6mm to less than 10mm, it has been classified by the previous studies as a "small polyp".

Their potential for advanced neoplasia is usually size-dependent, but some recent studies found that, even in diminutive and small polyps, the rate of advanced neoplasia is relatively high about 9%-10%.

The investigators will prospectively investigate postprocedural outcomes, such as retrieval rate, procedural time, overall complication rate (Intraprocedural bleeding, postprocedural bleeding, and perforation) in colonoscopic polypectomy of small polyp between CSP and EMR.

ELIGIBILITY:
Inclusion Criteria:

* All those over the age of 20 years who agree informed consent and who have at least one polyp of eligible size (6-10 mm)

Exclusion Criteria:

* (1) patients taking anticoagulant therapy during the past 1 week of the procedure, (2) known coagulopathy, (3) history of liver cirrhosis, chronic kidney disease, malignancy, inflammatory bowel diseases or significant infectious disease, (4) American Society of Anesthesiology class III or more, and (5) pedunculated polyps and polyps with malignant feature.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-09 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
complete resection rate (CRR) | Up to 2 months

SECONDARY OUTCOMES:
incidence of complications (Intraprocedural bleeding, postprocedural bleeding, and perforation) | Up to 2 months
necessity of hemostasis (due to Intraprocedural bleeding or postprocedural bleeding) | Up to 2 months
Polyp retrieval rate | Up to 2 months
hospitalization period | Up to 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Sik Byeon, Doctor, Study Chair — Division of Gastroenterology, Department of Internal Medicine, University of Ulsan College of Medicine, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Seoul, South Korea